CLINICAL TRIAL: NCT04828330
Title: Effects of Physical Activities on Pain and Functional Recovery in Low Back Pain
Brief Title: Flares of Low Back Pain With Activity Research Study
Acronym: FLAReS
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F3248-R; I01RX003248 (NIH)
Record Dates: First submitted 2021-03-22; First posted 2021-04-02 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational cohort: This is a case-crossover study nested within a cohort study.

SUMMARY:
Low back pain (LBP) is the most common cause of disability worldwide. Although general activity is encouraged in the treatment of LBP, there is limited empirical information available on the specific types of activities that are beneficial or harmful for patients seen in primary care for LBP. This study will identify those physical activities with short-term (transient) effects on LBP exacerbations (or "flares" of LBP), as well as identifying the long-term (cumulative) effects of such activities on functional recovery.

DETAILED DESCRIPTION:
This research will use a novel approach to distinguish the short-term effects on LBP of physical activities from the long-term effects of such activities, by conducting a longitudinal case-crossover study nested within a cohort study. This design accounts for measured and unmeasured confounds by using each case as his/her own control- an entirely observational study that is analogous to a crossover experiment- capitalizing on modern mobile health and actigraphy technology. The primary exposures of interest are 10 self-reported physical activities commonly performed during work and activities of daily living, and actigraphy-assessed physical activity. Other exposures of interest include psychological factors, social factors, lifestyle-related factors, and work-related factors. The primary outcomes are participant-reported "flares" of low back pain (Aim 1) and participant-reported back-related functional limitations (mobility and activities of daily living [ADLs]) at 1-year follow-up, as measured by the Roland-Morris Disability Questionnaire. This observational study will include up to 550 Veterans with LBP aged 18 and older recruited from the VA Puget Sound Health Care System (VAPSHCS). The study will not affect participants' medical care in any way. After informed consent, recruitment, and baseline data collection, study participants will complete frequent, serial electronic "e-Questionnaires" using their own personal electronic devices (personal computer [PC], tablet, or smartphone) over the 1-year period of follow-up. Participants may also wear ActiGraph units for the 1st 4 weeks of follow-up. Long-term outcomes will be assessed by extended e-Questionnaires completed at 1-year follow-up. Aim 1 analyses will examine the short-term effects of 10 specific activity categories on participant-reported flares across all study assessments over 1-year follow-up. Aim 2 analyses will examine associations between the frequency of exposure to 10 specific activity categories over weeks 1-4 of follow-up, and long-term functional recovery at 12 months as defined by the RMDQ. All analyses will use a biopsychosocial framework accounting for potential confounders (sociodemographics, psychological factors, etc.) and effect modifiers, and will include sensitivity analyses to examine the robustness of findings and important study assumptions. This study was registered prior to the start of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age 18-65 years seen in VA primary care for LBP
* Must have regular access (every day, during most hours of the day) to a computer, tablet, or smartphone with internet access at home or at work
* Basic computer literacy
* Having a mobile phone capable of receiving alerts using text messages
* Must be able to understand and read English, sufficient to provide informed consent and validly complete the study assessments.
* Participants must complete basic requirements during a 2-week run-in period, such as completing e-Questionnaires

After approval by the study sponsor and IRB, an additional inclusion criterion was added beginning on 3/10/2023, to also allow the inclusion of other patients with low back pain. The inclusion criteria were broadened to include other patients seen for low back pain in the health care system, including three "specific" subgroups of Veterans with low back pain: (1) Veterans with lumbosacral facet-mediated low back pain; (2) Veterans with sacroiliac joint-mediated low back pain; and (3) Veterans with spondylolytic spondylolistheses.

Exclusion Criteria:

* Red flag' spine conditions (spinal cord injury, infection, malignancy, fracture) or spondyloarthropathy
* Pregnancy
* Prisoners or incarcerated
* Severe active medical or psychiatric comorbidities likely to be a barrier to study participation including completing frequent, serial assessments (e.g., metastatic cancer).
* Thoracolumbar spine surgery in the past 1 year
* Other major orthopedic surgery potentially impeding normal physical activities (such as surgeries involving the hip, knee, ankle, shoulder, elbow, wrist joints) within the past 6 months, or major abdominal or chest surgery within the past 6 months.*
* Planned major orthopedic, abdominal, or chest surgery in the next 2 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans age 18-65 years seen in VA primary care for LBP
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Suri, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Only completely deidentified/anonymized versions of datasets would be shared, provided that appropriate VA enterprise-level procedures permit this and are in place at the time of. These procedures do not currently exist but are expected in the future. Sharing would only take place under a written agreement prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset, and would require a properly submitted FOIA request. Due to the project's waiver of HIPAA authorization, a subset of the data cannot be disclosed to a non-Federal entity. Electronic versions of final data sets will be maintained locally in a secure manner until enterprise-level resources become available for long-term storage.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will endeavor to be able to share IPD when requested by 6 months after the time of publication of the main study findings and publication of longer-term results of the study, provided that appropriate enterprise-level procedures permit this and are in place at the time of.
Access Criteria: The study team and PI will review each request for IPD, with involvement of local administrative officials or ORD officials as appropriate. Requests will be evaluated for criteria including data safety, the purpose of analyses warranting potential risks of transferring data, security of the transfer. An agreement will specify the duration of time for data to be held before

REFERENCES:
- [Background] Suri P, Tanus AD, Torres N, Timmons A, Irimia B, Friedly JL, Korpak A, Daniels C, Morelli D, Hodges PW, Costa N, Day MA, Heagerty PJ, Jensen MP. The Flares of Low back pain with Activity Research Study (FLAReS): study protocol for a case-crossover study nested within a cohort study. BMC Musculoskelet Disord. 2022 Apr 21;23(1):376. doi: 10.1186/s12891-022-05281-1. PMID 35449043

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational Cohort
Started | 416
Completed | 416
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Observational Cohort
Number analyzed (Participants) | 416
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years
  years | 47.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 6 participants had missing data for sex
  Participants
    number analyzed (Participants) | 410
    Female | 306
    Male | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52
  Not Hispanic or Latino | 328
  Unknown or Not Reported | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 54
  White | 279
  More than one race | 35
  Unknown or Not Reported | 18
Roland-Morris Disability Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Roland-Morris Disability Questionnaire (RMDQ) is a back-specific measure of functional limitations ranging from 0 to 24, where 0 reflects no disability and 24 reflects severe disability.
  units on a scale | 12.2 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Participant-reported "Flares" of Low Back Pain (Aim 1)
Description: At each study assessment, participants are presented with the flare definition used in this study, which was derived from a previously validated flare definition by Costa et al (2000). The definition is: "A 'flare' of low back pain is a worsening of your low back pain that lasts from hours to weeks".
  Participants are then asked to self-report whether a flare of low back pain is currently ongoing, by responding to the question "According to the definition above, are you currently experiencing a flare of your low back pain?", with response options of "yes" or "no". These response options define participant-reported flares.
Time Frame: Flares over 1-year follow-up
Measure: Mean (Standard Deviation); unit: Mean flares per year
Arm/Group | Observational Cohort
Number analyzed (Participants) | 416
Mean flares per year | 7.3 (7.3)

2. Primary Outcome: Roland-Morris Disability Questionnaire (Aim 2)
Description: Roland-Morris Disability Questionnaire (RMDQ) is a back-specific measure of functional limitations ranging from 0 to 24, where 0 reflects no disability and 24 reflects severe disability.
Time Frame: 1-year follow-up
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Observational Cohort
Number analyzed (Participants) | 416
Units on a scale | 10.0 (6.3)

ADVERSE EVENTS:
Description: This was a purely observational study and not a randomized trial. No adverse event data were collected; the plan to not monitor adverse event data was approved in our IRB review process.
Arm/Group | Observational Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This was a purely observational study. It was not a randomized trial. Due to the purely observational nature of the study, no adverse event data is provided, as no adverse event monitoring was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT04828330/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT04828330/ICF_000.pdf